CLINICAL TRIAL: NCT03627546
Title: A Randomized Study of a Rapid HCV Treatment Initiation Strategy (HCV Seek, Test and Rapid Treatment) Compared to Standard Care in Young People Who Inject Drugs
Brief Title: HCV Seek, Test and Rapid Treatment for Young PWID
Acronym: HCV ST&RT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1710018606
Record Dates: First submitted 2018-07-20; First posted 2018-08-13 (Actual); Results first posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2023-11

CONDITIONS: Hepatitis C; Drug Use
Keywords: PWID
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Rapid Treatment with sofosbuvir/velpatasvir (Intervention arm) (Experimental): The intervention arm receives same-day medical evaluation and treatment for hepatitis C. They receive medical evaluation, laboratory assessment , baseline questionnaire/interview, and distribution of a medication (sofosbuvir/velpatasvir) "starter pack" on the day of enrollment. Participants who are HCV RNA negative are followed separately and do not receive intervention. Other participants start medications and receive weekly text messages during treatment to record adherence. They have follow up visits for laboratory tests, medication distribution, and counseling for prevention of reinfection. They have HCV testing at end of treatment and 12 weeks post treatment, and at 48 weeks to assess for reinfection. Each study visit will include a brief questionnaire and qualitative interview.
  Interventions: Other: Rapid Treatment strategy
- Usual Care (Control arm) (Active Comparator): Participants in the control arm will be provided facilitated referral to community HCV providers by an on-site care coordinator already facilitating care at the community site. HCV RNA negative participants will be called to inform them of these results, and then followed separately. HCV RNA positive participants will be asked during the semi-structured interviews as at 12, 24, 36 and 48 week if they engaged in HCV treatment to assess whether their HCV referral has been filled, and to record their current HCV treatment status. They will also receive repeat HCV RNA testing at week 12, 24, and 48. Participants that have started treatment will be asked to sign consent for release of medical records pertaining to HCV-related laboratory testing to determine achievement of treatment response.
  Interventions: Other: Usual Care (facilitated referral)
- HCV RNA negative (No Intervention): Participants assigned to either group who were found to be HCV RNA-negative at entry. They are not eligible for treatment and thus not part of the analysis. They were asked to return the treatment starter pack. They are followed with HCV RNA measured at Week 24 and 48.

INTERVENTIONS:
Other: Rapid Treatment strategy — The intervention arm receives same-day medical evaluation and treatment for hepatitis C. They receive medical evaluation, laboratory assessment , baseline questionnaire/interview, and distribution of a medication (sofosbuvir/velpatasvir) "starter pack" on the day of enrollment. Participants who are HCV RNA negative are discontinued from the study. Other participants start medications and receive weekly text messages during 12 weeks of provided sofusbuvir/velpatasvir treatment.
  Arms: Rapid Treatment with sofosbuvir/velpatasvir (Intervention arm)
Other: Usual Care (facilitated referral) — articipants in the control arm will be provided facilitated referral to community HCV providers by an on-site care coordinator already facilitating care at the community site. HCV RNA negative participants will be called to inform them of these results, and then followed separately. HCV RNA positive participants will be asked during the semi-structured interviews as at 12, 24, 36 and 48 week if they engaged in HCV treatment to assess whether their HCV referral has been filled, and to record their current HCV treatment status. They will also receive repeat HCV RNA testing at week 12, 24, and 48. Participants that have started treatment will be asked to sign consent for release of medical records pertaining to HCV-related laboratory testing to determine achievement of treatment response.
  Arms: Usual Care (Control arm)

SUMMARY:
The purpose of this randomized study is to determine whether a community-based test and treat model of hepatitis C (HCV) care delivery will be superior to the usual care practice of referral to specialist clinics for the outcomes of sustained virologic response at 12 weeks after treatment and initiation of HCV treatment for persons who inject drugs (PWID) between ages 18 and 29 who are naïve to HCV treatment

DETAILED DESCRIPTION:
ST&RT is a randomized open-label clinical trial in which 54 HCV infected PWID between ages 18 and 29 will be randomized to either receive the same-day treatment initiation of the FDA-approved fixed dose combination of sofosbuvir 400mg and velpatasvir 100mg (SOF/VEL) with follow up and medical monitoring at a community site (Intervention arm) or to receive referral to an HCV treatment provider's office (Usual Care Arm).

ELIGIBILITY:
Inclusion Criteria:

* Persons are eligible for study inclusion if they: (a) are HCV antibody positive, (b) are 18 to 29 years of age, (c) have injected drugs in the past 30 days, (d) are HCV treatment naïve, (e) are English speaking

Exclusion Criteria:

* Persons excluded from the study will be (a) HIV coinfected persons (b) pregnant women, or women planning on becoming pregnant (c) participants with end-stage renal disease (d) participants with decompensated cirrhosis (c) participants on medications with treatment limiting interactions with sofosbuvir/velpatasvir

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Marks, Principal Investigator — Weill Cornell MC
Locations (1):
- Lower East Side Harm Reduction Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Baseline RNA-positive Rapid Treatment With Sofosbuvir/Velpatasvir (Intervention Arm): The intervention arm receives same-day medical evaluation and treatment for hepatitis C. They receive medical evaluation, laboratory assessment , baseline questionnaire/interview, and distribution of a medication (sofosbuvir/velpatasvir) "starter pack" on the day of enrollment. Participants who are HCV RNA negative are discontinued from the study. Other participants start medications and receive weekly text messages during treatment to record adherence. They have follow up visits for laboratory tests, medication distribution, and counseling for prevention of reinfection. They have HCV testing at end of treatment and 12 weeks post treatment, and at 48 weeks to assess for reinfection. Each study visit will include a brief questionnaire and qualitative interview.
  Sofosbuvir and Velpatasvir: Sofosbuvir/velpatasvir (Epclusa) is an FDA-approved treatment for HCV. It is provided in the intervention arm as part of a rapid treatment strategy,
- Baseline RNA-positive Usual Care (Control Arm): Participants in the control arm will be provided facilitated referral to community HCV providers by an on-site care coordinator already facilitating care at the community site. HCV RNA negative participants will be called to inform them of these results, and then discontinued from the study. HCV RNA positive participants will be asked during the semi-structured interviews as at 12, 24, 36 and 48 week if they engaged in HCV treatment to assess whether their HCV referral has been filled, and to record their current HCV treatment status. They will also receive repeat HCV RNA testing at week 12, 24, and 48. Participants that have started treatment will be asked to sign consent for release of medical records pertaining to HCV-related laboratory testing to determine achievement of treatment response.
- Baseline RNA Negative: Participants assigned to either group who were found to be HCV RNA-negative at entry. They are not eligible for treatment and thus not part of the analysis. They were asked to return the treatment starter pack. They are followed with HCV RNA measured at Week 24 and 48.
Period: Overall Study
Arm/Group | Baseline RNA-positive Rapid Treatment With Sofosbuvir/Velpatasvir (Intervention Arm) | Baseline RNA-positive Usual Care (Control Arm) | Baseline RNA Negative
Started | 15 | 11 | 13
Completed | 14 | 11 | 0
Not Completed | 1 | 0 | 13
Not completed — Deemed ineligible after ransdomization | 1 | 0 | 0
Not completed — HCV RNA Negative (protocol pre-specified) | 0 | 0 | 13

BASELINE CHARACTERISTICS:
Population: One participant was deemed ineligible after randomization and is not included. Participants found to be RNA negative at baseline are listed separately since they do not have hepatitis C infection and are not eligible for treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Baseline RNA-positive Rapid Treatment With Sofosbuvir/Velpatasvir (Intervention Arm) | Baseline RNA-positive Usual Care (Control Arm) | Baseline RNA Negative | Total
Number analyzed (Participants) | 14 | 11 | 13 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.07 (3.54) | 25.36 (2.66) | 26.92 (2.87) | 26.16 (3.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 10
  Male | 11 | 8 | 9 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Non-Hispanic White | 6 | 6 | 9 | 21
  Race/ethnicity: Non-Hispanic Black | 1 | 0 | 0 | 1
  Race/ethnicity: Hispanic | 6 | 3 | 4 | 13
  Race/ethnicity: Other | 1 | 2 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 14 | 11 | 13 | 38

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Participants Who Achieve Sustained Virologic Response 12 (SVR12) With Rapid Treatment Strategy Compared to Usual Care
Description: The proportion of participants who achieve sustained virologic response defined as an undetectable HCV RNA viral load 12 weeks after the cessation of treatment (SVR12), in the intervention arm compared to the usual care arm by study week 48.
Time Frame: Week 48
Population: Thirteen participants who were HCV-RNA negative at baseline excluded from analysis since they do not have hepatitis C and are not eligible for treatment. One participant in the intervention arm was deemed ineligible after randomization and was not included in analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Rapid Treatment With Sofosbuvir/Velpatasvir (Intervention Arm): The intervention arm receives same-day medical evaluation and treatment for hepatitis C. They receive medical evaluation, laboratory assessment , baseline questionnaire/interview, and distribution of a medication (sofosbuvir/velpatasvir) "starter pack" on the day of enrollment. Participants who are HCV RNA negative are discontinued from the study. Other participants start medications and receive weekly text messages during treatment to record adherence. They have follow up visits for laboratory tests, medication distribution, and counseling for prevention of reinfection. They have HCV testing at end of treatment and 12 weeks post treatment, and at 48 weeks to assess for reinfection. Each study visit will include a brief questionnaire and qualitative interview.
  Sofosbuvir and Velpatasvir: Sofosbuvir/velpatasvir (Epclusa) is an FDA-approved treatment for HCV. It is provided in the intervention arm as part of a rapid treatment strategy,
- Usual Care (Control Arm): Participants in the control arm will be provided facilitated referral to community HCV providers by an on-site care coordinator already facilitating care at the community site. HCV RNA negative participants will be called to inform them of these results, and then discontinued from the study. HCV RNA positive participants will be asked during the semi-structured interviews as at 12, 24, 36 and 48 week if they engaged in HCV treatment to assess whether their HCV referral has been filled, and to record their current HCV treatment status. They will also receive repeat HCV RNA testing at week 12, 24, and 48. Participants that have started treatment will be asked to sign consent for release of medical records pertaining to HCV-related laboratory testing to determine achievement of treatment response.
Arm/Group | Rapid Treatment With Sofosbuvir/Velpatasvir (Intervention Arm) | Usual Care (Control Arm)
Number analyzed (Participants) | 14 | 11
Participants | 9 | 1
Statistical Analysis 1: Comparison: Rapid Treatment With Sofosbuvir/Velpatasvir (Intervention Arm) vs Usual Care (Control Arm); Test type: Superiority; p = .01, Chi-squared

2. Secondary Outcome: The Proportion of Participants Who Initiate Treatment for HCV
Description: The proportion of participants who initiate treatment for HCV in the intervention arm compared to the usual care arm by study week 48.
Time Frame: Week 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rapid Treatment With Sofosbuvir/Velpatasvir (Intervention Arm) | Usual Care (Control Arm)
Number analyzed (Participants) | 14 | 11
Participants | 13 | 3
Statistical Analysis 1: Comparison: Rapid Treatment With Sofosbuvir/Velpatasvir (Intervention Arm) vs Usual Care (Control Arm); Test type: Superiority; p = 0.0007, Chi-squared

3. Secondary Outcome: Presence of Resistance Associated Substitutions (RAS) in Treated Patients With Treatment Failure
Time Frame: 48 wks
Population: Resistance testing data was not collected.
Arm/Group | Rapid Treatment With Sofosbuvir/Velpatasvir (Intervention Arm) | Usual Care (Control Arm)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants in Both Arms Who Achieve SVR12, or Are RNA Negative at Baseline, That Have HCV Reinfection by Study Week 48
Time Frame: 48 wks
Measure: Count of Participants; unit: Participants
Arm/Group | Rapid Treatment With Sofosbuvir/Velpatasvir (Intervention Arm) | Usual Care (Control Arm) | Baseline RNA Negative
Number analyzed (Participants) | 14 | 11 | 13
Participants | 1 | 0 | 1

5. Secondary Outcome: Impact of Engagement in HCV Treatment on Frequency of Substance Use or Injection Risk Behaviors
Description: Change in substance use frequency or injection risk behaviors will be defined as percent of participants in each arm that injected alone and the percent of participants who injected with 3 or more individuals
Time Frame: Baseline and 48 weeks
Population: Thirteen participants who were HCV-RNA negative at baseline excluded from analysis since they do not have hepatitis C and are not eligible for treatment. Not all participants completed the survey at Week 48.
Measure: Count of Participants; unit: Participants
Arm/Group | Rapid Treatment With Sofosbuvir/Velpatasvir (Intervention Arm) | Usual Care (Control Arm)
Number analyzed (Participants) | 14 | 11
Participants
  Entry: Injected with 3 or more individuals | 3 | 2
  Entry: Injected with 1-2 indivuduals | 10 | 5
  Entry: Injected alone | 1 | 4
  Entry: Did not inject | 0 | 0
  Week 48: number analyzed (Participants) | 10 | 7
  Week 48: Injected with 3 or more individuals | 1 | 1
  Week 48: Injected with 1-2 indivuduals | 3 | 4
  Week 48: Injected alone | 1 | 0
  Week 48: Did not inject | 5 | 2

ADVERSE EVENTS:
Time Frame: 12 months
Description: Thirteen participants who were HCV-RNA negative at baseline excluded from analysis since they do not have hepatitis C and are not eligible for treatment. One participant in the intervention arm was deemed ineligible after randomization and was not included in analysis. All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed in the "Baseline RNA Negative" Arm/Group
Groups:
- Baseline RNA Negative: Participants assigned to either group who were found to be HCV RNA-negative at entry. They are not eligible for treatment and thus not part of the analysis. They were asked to return the treatment starter pack. They are followed with HCV RNA measured at Week 24 and 48. All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed in the "Baseline RNA Negative" Arm/Group
Arm/Group | Rapid Treatment With Sofosbuvir/Velpatasvir (Intervention Arm) | Usual Care (Control Arm) | Baseline RNA Negative
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/11 | 0/0
Serious Adverse Events (participants affected / at risk) | 6/14 | 5/11 | 0/0
Other Adverse Events (participants affected / at risk) | 0/14 | 0/11 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rapid Treatment With Sofosbuvir/Velpatasvir (Intervention Arm) (N=14) | Usual Care (Control Arm) (N=11) | Baseline RNA Negative (N=0)
Drug overdose (Injury, poisoning and procedural complications) | 2 (2) | 4 (6) | 0
Skin/soft tissue infection (Infections and infestations) | 3 (3) | 0 (0) | 0
pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0
miscarriage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0
Spleen laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0
Seizure from withdrawal (Nervous system disorders) | 0 (0) | 1 (2) | 0
GI bleed (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT03627546/Prot_SAP_000.pdf